CLINICAL TRIAL: NCT05811364
Title: The GORE VBX FORWARD Clinical Study: A Comparison of the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis to Bare Metal Stenting for Patients With Complex Iliac Occlusive Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VBX 22-06
Record Dates: First submitted 2023-03-14; First posted 2023-04-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Aortoiliac Occlusive Disease; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Subject randomized to a VBX device group and BMS control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Every effort will be made to blind subjects to the treatment device up to the 1 year follow up visit. The independent Core Lab and Clinical Events Committee (CEC) members will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- VBX Device Group (Active Comparator): Subject in this group will receive treatment with the GORE VIABAHN® VBX Balloon Expandable Endoprosthesis (VBX)
  Interventions: Device: Stenting of the Common and/or External Iliac Arteries with the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis
- BMS Control Group (Active Comparator): Subjects in this group will receive treatment with a commercially available bare metal stent (BMS) that is approved for treatment of the disease
  Interventions: Device: Stenting of the Common and/or External Iliac Arteries with Bare Metal Stent

INTERVENTIONS:
Device: Stenting of the Common and/or External Iliac Arteries with the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis — Treatment of target lesions in the common and/or external iliac arteries by stenting with the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis.
  Arms: VBX Device Group
Device: Stenting of the Common and/or External Iliac Arteries with Bare Metal Stent — Treatment of target lesions in the common and/or external iliac arteries by stenting with a commercially available bare metal stent that is approved for treatment of the disease.
  Arms: BMS Control Group

SUMMARY:
The objective of this prospective, multicenter, randomized, controlled clinical trial is to demonstrate the superiority of the VBX Device for primary patency when compared to bare metal stenting in complex iliac occlusive disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of informed consent signature
* Informed Consent Form (ICF) is signed by the subject
* Subject can comply with protocol requirements, including follow-up
* Patient has symptomatic claudication, rest pain, or minor tissue loss (Rutherford Category 2-5)
* Patient has de novo or restenotic lesion(s) found in the common and/or external iliac artery(ies)
* Patient has: Unilateral or bilateral single or multiple lesions (>50% stenosis or chronic total occlusion) each between 4 and 11 cm in length
* Patient has a target vessel diameter visually estimated to be approximately between 5 mm and 13 mm
* Patient has a sufficient (<50% stenotic) common femoral artery and at least one sufficient (<50% stenotic) femoral artery (deep or superficial).
* Patient has at least one sufficient (<50% stenotic) infrapopliteal run-off vessel.

Exclusion Criteria:

* Life expectancy <1 year
* Patient is pregnant at time of informed consent.
* Patient has a known allergy to stent or stent graft components (including nitinol, stainless steel, or heparin).
* Patient has severe chronic renal insufficiency (serum creatinine level > 2.5mg/dL) and not undergoing hemodialysis.
* Patient has evidence of a systemic infection.
* Patient has a known intolerance to antithrombotic medications that prevent compliance with study or control device Instructions for Use.
* Patient has had vascular catheterization of the lower extremities within 30 days of randomization (excluding diagnostic angiograms for the study procedure).
* Patient has previous stenting in the iliac arteries.
* Patient has previous surgical bypass in the target limb.
* Patient is currently participating in another investigative clinical study unless received written approval by the sponsor.
* Patient has a lesion requiring drug-coated balloon angioplasty, atherectomy, lithotripsy, or any ablative device to facilitate stent delivery.
* Patient has an abdominal aortic artery lesion or aneurysm.
* Patient has a lesion that requires stent placement within 2 cm of the inguinal ligament.
* Patient has isolated common iliac artery stenosis that can be treated with a single device (i.e., common iliac artery stenosis that does not require kissing stents or extend into the external iliac artery).
* Patient has outflow disease that requires concomitant interventions (i.e. common femoral endarterectomy or femoral / tibial revascularization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary Patency | 1 year
  Blood flow through the target lesion (no evidence of binary restenosis >50% or occlusion) without a Target Lesion Revascularization (TLR).

SECONDARY OUTCOMES:
Technical success | at the procedure
  Deployment of device with < 30% residual stenosis on final angiography.
Acute procedural success | at the procedure
  Binary assessment based on technical success and freedom from device or procedure-related serious adverse events (SAE) requiring intervention.
Clinical success | Through 1 month
  Improvement from baseline of at least 1 Rutherford Category and freedom from device or procedure-related SAE requiring intervention.
Hemodynamic Status | Through 5 years
  Change in Ankle-brachial index (ABI)/toe-brachial index (TBI) as compared to baseline
Change in EQ-5D-5L | Through 5 years
  Change in EQ-5D-5L responses as compared to baseline. The EQ-5D-5L Questionnaire measures quality of life (QoL) over 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is measured over five levels from no problems to extreme problems. Scored on a 0 to 100 scale with 0 as the worst possible health and 100 is the best possible health.
Change in WIQ | Through 5 years
  Change in Walking Impairment Questionnaire (WIQ) responses as compared to baseline. The WIQ is a validated QoL measurement of walking abilities over 3 dimensions: distance, speed, and stair-climbing. Scored on a 0 to 100 scale with 0 as no degree of difficulty and 100 is the highest degree of difficulty.
Primary patency | Through 5 years
  Blood flow through the target lesion (no evidence of binary restenosis >50% or occlusion) without a Target Lesion Revascularization (TLR).
Freedom from binary restenosis | Through 5 years
  Freedom from binary restenosis. binary restenosis defined as evidence of >50% restenosis or occlusion of the target lesion(s) based on core lab adjudicated duplex ultrasound or angiography
Primary assisted patency | Through 5 years
  Blood flow maintained (no evidence of occlusion) through the target lesion with or without a Target Lesion Revascularization (TLR).
Secondary patency | Through 5 years
  Blood flow through the target lesion with or without a Target Lesion Revascularization (TLR).
Freedom from target lesion revascularization | Through 5 years
  Freedom from target lesion revascularization (TLR). TLR defined as endovascular or surgical intervention performed on the target lesion(s).
Cumulative reintervention rate | Through 5 years
  Rate of first and recurrent Target Lesion Revascularization (TLR).
Freedom from clinically driven target lesion revascularization | Through 5 years
  Freedom from clinically driven target lesion revascularization. Endovascular or surgical intervention performed on the target lesion(s) in response to recurrent symptoms (increase ≥ 1 Rutherford Category).
Amputation-free survival | Through 5 years
  Binary assessment based on freedom from major amputation (target limb, amputation above the metatarsals) and all-cause mortality
Survival | Through 5 years
  Freedom from all-cause mortality
Change in Rutherford Category | Through 5 years
  Change in Rutherford Category as compared to baseline. Scaled from 0 to 6, with 0 as asymptotic and 6 as major tissue loss, extending above the transmetatarsal (TM) level, functional foot no longer salvageable.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - North Suburban Medical Center, Denver, Colorado
  - Radiology and Imaging Specialists of Lakeland, Lakeland, Florida
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
- Krankenhaus der Barmherzigen Brüder, Regensburg, Germany
- Rijnstate Hospital, Arnhem, Netherlands
- Auckland City Hospital, Auckland, New Zealand

REFERENCES:
- [Derived] Kirkwood ML, Armstrong EJ, Ansari MM, Holden A, Reijnen MMPJ, Steinbauer M, Crannell Z, Novoa H, Phillips A, Schneider DB. FORWARD Study of GORE VIABAHN Balloon-Expandable Endoprostheses and Bare Metal Stents in the United States, European Union, United Kingdom, Australia, and New Zealand When Placed to Treat Complex Iliac Occlusive Disease: Protocol for a Randomized Superiority Trial. JMIR Res Protoc. 2023 Dec 4;12:e51480. doi: 10.2196/51480. PMID 38048145